CLINICAL TRIAL: NCT03528434
Title: for Infection Prevention in Sickle Cell Anemia (ZIPS)
Brief Title: Zinc for Infection Prevention in Sickle Cell Anemia (ZIPS)
Acronym: ZIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Makerere University (Other); Jinja Regional Referral Hospital (Unknown); Université de Montréal (Other)
Responsible Party: Principal Investigator, Chandy John, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1712339562
Record Dates: First submitted 2018-05-07; First posted 2018-05-17 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Sickle Cell Disease
Keywords: Zinc
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Zinc

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, double blind clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc (Experimental): Dietary Supplement: Zinc 10mg dispersible zinc sulfate tablet
  Interventions: Dietary Supplement: Zinc
- Placebo (Placebo Comparator): Dispersible tablet with inert ingredients, identical to zinc in appearance
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc — 10mg dispersible zinc sulfate tablet
  Arms: Zinc
Other: Placebo — Dispersible tablet with inert ingredients, identical to zinc in appearance
  Arms: Placebo

SUMMARY:
A randomized double-blinded placebo-controlled trial of zinc to reduce the incidence of severe or invasive infections in Ugandan children with sickle cell anemia (SCA).

DETAILED DESCRIPTION:
The study will be a randomized, placebo-controlled, double blind clinical trial in which 250 Ugandan children 1.00-4.99 years of age with SCA will receive zinc (10 mg oral dispersible tablet daily) or placebo (identical to zinc in appearance) for 12 months. The primary study outcome will be incidence of severe or invasive infections. Secondary outcomes will include incidence of all clinical infections, confirmed bacterial infections (by culture or PCR), incidence of vaso-occlusive crisis (VOC), change in height-for-age z-score, and incidence of zinc-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Documented sickle cell anemia (HbSS supported by hemoglobin electrophoresis)
2. Age range of 1.00-4.99 years, inclusive, at the time of enrollment
3. Weight at least 5.0 kg at the time of enrollment
4. Willingness to comply with all study-related treatments, evaluations, and follow-up

Exclusion Criteria:

1. Known other chronic medical condition (e.g., HIV, malignancy, active clinical tuberculosis)
2. Severe malnutrition determined by impaired growth parameters as defined by the World Health Organization (WHO) (weight for length/height or height for age z-score <-3, using WHO growth standards)

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Incidence of infection | 12 months
  The investigators will assess reduction in incidence of severe or invasive infections, with or without culture or PCR confirmation.

SECONDARY OUTCOMES:
Incidence of all clinical infections | 12 months
  Incidence of all clinical infections
Incidence of confirmed bacterial infections (by culture or PCR) | 12 months
  Incidence of confirmed bacterial infections (by culture or PCR)
Incidence of vaso-occlusive crisis (VOC) | 12 months
  Incidence of vaso-occlusive crisis (VOC)
Change in height-for-age z-score | Enrollment to 12 months
  Change in height-for-age z-score
Incidence of zinc-related adverse events | 12 months
  Incidence of zinc-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chandy C. John, MD, Principal Investigator — Indiana University
Locations (1):
- Jinja Reginal Referral Hospital, Jinja, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bolarinwa AB, Oduwole O, Okebe J, Ogbenna AA, Otokiti OE, Olatinwo AT. Antioxidant supplementation for sickle cell disease. Cochrane Database Syst Rev. 2024 May 22;5(5):CD013590. doi: 10.1002/14651858.CD013590.pub2. PMID 38775255
- [Derived] Namazzi R, Opoka R, Conroy AL, Datta D, Tagoola A, Bond C, Goings MJ, Ryu MS, Cusick SE, Krebs NF, Jang JH, Tu W, Ware RE, John CC. Zinc for infection prevention in children with sickle cell anemia: a randomized double-blind placebo-controlled trial. Blood Adv. 2023 Jul 11;7(13):3023-3031. doi: 10.1182/bloodadvances.2022008539. PMID 36735400
- [Derived] Datta D, Namazzi R, Conroy AL, Cusick SE, Hume HA, Tagoola A, Ware RE, Opoka RO, John CC. Zinc for Infection Prevention in Sickle Cell Anemia (ZIPS): study protocol for a randomized placebo-controlled trial in Ugandan children with sickle cell anemia. Trials. 2019 Jul 26;20(1):460. doi: 10.1186/s13063-019-3569-z. PMID 31349866

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT03528434/Prot_SAP_000.pdf